CLINICAL TRIAL: NCT00242190
Title: Gemcitabine, Oxaliplatin and Radiation Therapy in Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2003-082
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Pancreatic Neoplasms
Keywords: drug therapy; radiotherapy; clinical trial
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Gemcitabine; Radiotherapy

INTERVENTIONS:
Drug: oxaliplatin
Drug: gemcitabine
Procedure: radiation therapy

SUMMARY:
This study will examine a proposed research treatment which evaluates the addition of oxaliplatin, a chemotherapy agent, to gemcitabine, another chemotherapy agent, and radiation therapy for the treatment of patients with pancreatic cancer. The researchers have already done studies using gemcitabine and radiation therapy together. They want to build on the information they have from this previous research. The researchers believe that the combination chemotherapy with radiation is worth investigating to treat pancreatic cancer. They will use this study to determine what type of side effects occur with this treatment and to assess how effective the treatment is at controlling the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologic or histologic confirmation of carcinoma arising in the pancreas.
* Patients may have any stage of pancreatic cancer but if metastatic, systemic disease burden should be asymptomatic and small in volume.
* Determination of resectability must be made prior to registration.
* Patients must have an estimated life expectancy of at least 12 weeks and a Zubrod performance status of < = 2.
* Patients must have adequate organ function defined as follows: absolute neutrophil count of > = 1500/mm3, platelets > = 100,000/mm3, serum Cr < = 1.5 mg/dl, bilirubin < 3.0 mg/dl, with relief of biliary obstruction if present (PTC tube or endobiliary stent).
* Patients must be free of other active systemic malignancy, ongoing infection, including HIV infection, or any other serious uncontrolled, concomitant systemic disorders or psychiatric condition that would interfere with the safe delivery of protocol therapy.
* Patients of reproductive potential must have agreed to use an effective contraceptive method during participation in this trial and for 6 months after trial.
* Patient must be aware of the investigational nature of the therapy and provide written informed consent.

Exclusion Criteria:

* Patients with neuroendocrine tumors are excluded.
* Patients must have no history of previous chemotherapy for pancreatic cancer or any abdominal radiation therapy.
* Patient must not have used any investigational agent in the month before enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-06; Primary Completion 2006-03 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicity up to three weeks following the second cycle of chemotherapy.

SECONDARY OUTCOMES:
Characterize pattern of responses, progression free survival, and survival after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States